CLINICAL TRIAL: NCT00283231
Title: RESPeRATE (Paced Respiration) for Treatment of Hot Flashes and Menopausal Symptoms
Brief Title: RESPeRATE for Treatment of Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H5287-27101
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2005-07

CONDITIONS: Menopause
Keywords: Hot Flashes; Menopausal Symptoms; Paced respiration; RESPeRATE
MeSH Terms: conditions — Hot Flashes

INTERVENTIONS:
Behavioral: Paced Respiration

SUMMARY:
This is an uncontrolled pilot clinical trial to determine the feasibility of recruitment and effectiveness of a device called RESPeRATE that paces respiration to treat menopausal hot flashes in 12 peri- or postmenopausal women. Participants will practice paced respiration for 15 minutes everyday for six weeks and attend assessment visits at weeks 3 and 6.

DETAILED DESCRIPTION:
This is an uncontrolled pilot trial of the effects of learning paced respiration using RESPeRATE in 12 healthy peri- or postmenopausal women between 40 and 60 years old who report experiencing at least 4 hot flashes per day or 30 hot flashes per week. Participants will be screened by telephone, then attend a clinic visit for further screening, and a baseline visit for final eligibility assessment and to learn how to use the RESPeRATE. Participants will receive information about the use of the RESPeRATE and paced respiration from a trained staff member and practice using the RESPeRATE during the clinic visit. Participants will also be instructed how to record hot flashes in a diary. The intervention will consist of using the RESPeRATE device for 15 minutes daily. Outcomes will be assessed in the clinic after 3 weeks and 6 weeks use of the device. The main efficacy outcomes are change in number of hot flashes per week and change in hot flash score (number of flashes x mean severity) from baseline to 3 and 6 weeks post-training, reported on the 7-day diary. Frequency of hot flashes will also be measured at baseline and 6 weeks using a 24-hour ambulatory hot flash monitor. Change in breathing rate will be calculated from baseline to 3 and 6 weeks and changes in sleep and quality of life from baseline to 6 weeks as measured by validated self-administered questionnaires. The mechanism of response to the RESPeRATE will be explored by measuring blood pressure at baseline, 3 weeks and 6 weeks and, body mass index and 24-hour levels of urinary epinephrine, norepinephrine and cortisol at baseline and 6 weeks. We will also draw a fasting blood sample at baseline and 6 weeks to measure serum lipids, glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Self-report >4 hot flashes per day or ≥ 30 hot flashes per week.
2. Successful completion of a Hot Flash Diary.
3. Willingness to attend all visits, fast before blood draws, complete all questionnaires, complete the hot flash diary, wear an ambulatory monitor, collect a 24-hour urine and wear the RESPeRATE for 15 minutes per day.
4. Agree not to use therapies that may affect hot flashes during the trial (estrogens, progestins, raloxifene, tamoxifen, clonidine, selective serotonin reuptake inhibitors, relaxation techniques or acupuncture). -

Exclusion Criteria:

1. Inability to sign an informed consent or fill out questionnaires.
2. Use of therapies that may affect hot flashes within 4 weeks of entering the trial (estrogens, progestins, raloxifene, tamoxifen, clonidine, selective serotonin reuptake inhibitors, relaxation techniques or acupuncture).
3. History of pulmonary disease including emphysema, chronic bronchitis, or chronic obstructive pulmonary disease (COPD).
4. Pregnant or breast feeding.
5. Any condition that, in the investigator's opinion, would preclude the participant from being able to understand and use the RESPeRATE device or complete the trial, including severe illness, (e.g., active ischemic heart disease/unstable angina, severe congestive heart failure, chronic atrial fibrillation, stroke resulting in permanent impairment, chronic renal failure or sleep paralysis), plans to move, substance abuse, significant psychiatric problems, or dementia.
6. Blood pressure during screening of ≤ 100/60 mmHg.
7. Current use of any medication prescribed to lower blood pressure.

   -

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-10; Study Completion 2006-02

PRIMARY OUTCOMES:
The efficacy of the intervention for reduction of number and severity of hot flashes will be summarized by the sample averages, with 95% confidence intervals.
We will also perform a paired t-test of the baseline and post-treatment values.

SECONDARY OUTCOMES:
Feasibility will be measured by number of weeks required to enroll 12 participants and the cost of recruitment per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Grady, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Women's Health Clinical Research Center, San Francisco, California, United States